CLINICAL TRIAL: NCT01335542
Title: Analgesia After Total Knee Arthroplasty: Peri-Articular Injection Versus Epidural + Femoral Nerve Blockade
Acronym: PAI vs FNB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2012-056
Record Dates: First submitted 2011-04-08; First posted 2011-04-14 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Readiness to Discharge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural Pathway (PCEA+FNB) (Active Comparator)
  Interventions: Procedure: Epidural Pathway (PCEA+FNB)
- Peri-Articular Injection (Active Comparator)
  Interventions: Procedure: Peri-Articular Injection

INTERVENTIONS:
Procedure: Peri-Articular Injection — Pre-operative anesthesia/analgesia: meloxicam (7.5 or 15mg), dexamethasone (6mg) Anesthetic:: Combined Spinal-Epidural with 0.5% bupivacaine. IV sedation with midazolam, propofol Antiemetic: 20mg famotidine, 4mg ondansetron Postoperative pain management: hydromorphone/bupivacaine PCEA (4/4/10/20, initially). Meloxicam (7.5 or 15mg), Oxycodone/Acetaminophen (5/325 3hr PRN)
  Arms: Peri-Articular Injection
Procedure: Epidural Pathway (PCEA+FNB) — Pre-operative anesthesia/analgesia: meloxicam (7.5 or 15mg), extended release oxycodone (10mg or 20mg), dexamethasone (6mg), clonidine patch (100 mcg/24 hr) Anesthetic: Spinal with 0.5% bupivacaine, IV sedation with midazolam, propofol Antiemetic: 20mg famotidine, 4mg ondansetron Post-operative analgesia:Prilosec (20mg), Meloxicam (7.5mg or 15 mg PO), extended release oxycodone (10mg or 20mg), Oxycodone (5mg q 3 hr PRN), Acetaminophen (1000mg), ketorolac 15mg IV
  Arms: Epidural Pathway (PCEA+FNB)

SUMMARY:
There are 2 common ways to manage pain after total knee arthroplasty at our institution. Some patients receive an epidural analgesia, a femoral nerve block and pills for pain. More recently, some surgeons have replaced femoral nerve blockade with peri-articular injections. These patients receive a peri-articular injection (injection of pain medication around the knee), pills for pain and a pain patch on the skin. The purpose of this research project is to find out if one of these ways to treat pain is better than the other. The investigators will look at this question in many ways, but the main way is how long it takes for you to be judged ready for discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for primary bicompartmental total knee arthroplasty with a participating surgeon
* Age 18 to 85 years old
* Planned use of regional anesthesia
* Ability to follow study protocol
* Up to 15 degrees varus, up to 15 degrees flexion and up to 15 degrees valgus

Exclusion Criteria:

* Patients younger than 18 years old and older than 85
* Patients intending to receive general anesthesia
* Allergy or intolerance to one of the study medications
* Patients with an ASA of IV
* Patients with insulin-dependent diabetes
* Patients with hepatic (liver) failure
* Patients with chronic renal (kidney) failure
* Chronic opioid use (taking opioids for longer than 3 months)
* Patients with any prior major ipsilateral open knee surgery.
* Patients with flexion contracture of knee > 15 degrees
* Patients with varus deformity > 15 degrees
* Patients with valgus deformity > 15 degrees
* Patients with a contraindication to use of epinephrine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, M.D., Ph.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient in the local infiltration group was deemed ineligible due to a rheumatoid arthritis. Only 90 patients were randomized to the study.
Groups:
- Epidural Pathway: meloxicam (7.5 or 15mg), extended release oxycodone (10mg or 20mg), dexamethasone (6mg), clonidine patch (100 mcg/24 hr) Anesthetic: Spinal with 0.5% bupivacaine, IV sedation with midazolam, propofol Antiemetic: 20mg famotidine, 4mg ondansetron Post-operative analgesia:Prilosec (20mg), Meloxicam (7.5mg or 15 mg PO), extended release oxycodone (10mg or 20mg), Oxycodone (5mg q 3 hr PRN), Acetaminophen (1000mg), ketorolac 15mg IV
- Local Infiltration: meloxicam (7.5 or 15mg), dexamethasone (6mg) Anesthetic:: Combined Spinal-Epidural with 0.5% bupivacaine. IV sedation with midazolam, propofol Antiemetic: 20mg famotidine, 4mg ondansetron Postoperative pain management: hydromorphone/bupivacaine PCEA (4/4/10/20, initially). Meloxicam (7.5 or 15mg), Oxycodone/Acetaminophen (5/325 3hr PRN)
Period: Overall Study
Arm/Group | Epidural Pathway | Local Infiltration
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient in the local infiltration group was deemed ineligible due to a rheumatoid arthritis. The remaining 90 patients were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Pathway | Local Infiltration | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 67 [50 to 84] | 65 [49 to 81] | 66 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90
BMI [Number; unit: participants]
  Normal | 3 | 2 | 5
  Overweight | 19 | 20 | 39
  Obese | 21 | 20 | 41
  Morbidly Obese | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is Time Until a Patient is "Ready for Discharge."
Description: The primary outcome is time until a patient is "ready for discharge." Discharge criteria are:
  * PCA (if present) has been discontinued
  * Not experiencing moderate or severe nausea (within last 4 hours).
  * Solid food diet
  * Able to urinate (Foley catheter removed)
  * Pain: NRS <4.
  * Surgical wound dry
  * No acute medical problems
  * Physical Therapy Criteria
    * Independently transfer from supine to sit, from sitting to standing
    * Ambulate 40 ft. without assistance
    * Extension range of motion (< 10 degrees)
Time Frame: Participants will be followed for the duration of their hospital stay, an expected average of 3 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Epidural Pathway | Local Infiltration
Number analyzed (Participants) | 45 | 45
days | 3.2 [1.8 to 7.0] | 3.2 [1 to 14]

ADVERSE EVENTS:
Arm/Group | Epidural Pathway | Local Infiltration
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes